CLINICAL TRIAL: NCT06690359
Title: Evaluation of IM19 CAR-T Cell Therapy for IgA Nephropathy With Urinary Protein and Renal Dysfunction Safety and Efficacy of Patients With Primary Membranous Nephropathy and Those at Medium to High Risk Clinical Research
Brief Title: IM19 CAR-T Cell Therapy for IgA Nephropathy Patients and Membranous Nephropathy Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZMA02
Record Dates: First submitted 2024-11-05; First posted 2024-11-15 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: IgA Nephropathy; Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulonephritis, Membranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IgA nephropathy subjects with urinary protein and renal insufficiency (Experimental): The study plans to recruit 6 patients with IgA nephropathy accompanied by urinary protein and renal dysfunction, including 3 patients receiving a dose of 0.5 × 10 ^ 8 CAR-T cells and 3 patients receiving a dose of 1 × 10 ^ 8 CAR-T cells
  Interventions: Combination Product: IM19 chimeric antigen receptor T cell injection
- Primary membranous nephropathy (Experimental): Recruiting 6 patients with medium to high-risk PMN, including 3 patients receiving 0.5 × 10 ^ 8 CAR-T cell dose and 3 patients receiving 1 × 10 ^ 8 CAR-T cell dose, for corresponding doses of IM19 CAR-T cell infusion therapy
  Interventions: Combination Product: IM19 chimeric antigen receptor T cell injection

INTERVENTIONS:
Combination Product: IM19 chimeric antigen receptor T cell injection — IgA nephropathy:
  The investigators plan to recruit IgA nephropathy subjects with urinary protein and renal dysfunction who meet the inclusion and exclusion criteria. They will receive Beijing Zaimiao Biological IM19 CAR-T cell infusion therapy at doses of 0.5 × 10 ^ 8 and 1 × 10 ^ 8 CAR-T cells, with 3 subjects enrolled at each dose
  Primary membranous nephropathy:
  The investigators plan to recruit primary membranous nephropathy subjects who meet the inclusion and exclusion criteria and receive IM19CAR-T cell infusion therapy at doses of 0.5 × 10 ^ 8 and 1 × 10 ^ 8 CAR-T cells, with 3 subjects enrolled at each dose

SUMMARY:
IM19 CAR-T cell therapy for IgA nephropathy patients with urinary protein and renal dysfunction, as well as patients with intermediate to high-risk primary membranous nephropathy

DETAILED DESCRIPTION:
IgA nephropathy:

The investigators plan to recruit IgA nephropathy subjects with urinary protein and renal dysfunction who meet the inclusion and exclusion criteria. They will receive IM19 CAR-T cell infusion therapy at doses of 0.5 × 10 ^ 8 and 1 × 10 ^ 8 CAR-T cells, with 3 subjects enrolled at each dose. The investigators will evaluate the changes in urinary protein and eGFR relative to baseline values within 6 months of the first infusion, the rate of reaching the threshold, and the occurrence of adverse events related to IM19 CAR-T cell infusion within 28 days after the infusion.

And evaluate the long-term efficacy, namely the changes in urinary protein and eGFR relative to baseline values and the ratio of reaching threshold values after 360 days of cell transfusion. The retention amount and duration of IM19 CAR-T cells in the peripheral blood of subjects.

Primary membranous nephropathy:

The investigators plan to recruit primary membranous nephropathy subjects who meet the inclusion and exclusion criteria and receive IM19CAR-T cell infusion therapy at doses of 0.5 × 10 ^ 8 and 1 × 10 ^ 8 CAR-T cells. Three subjects will be enrolled at each dose to evaluate the changes and disappearance rate of PLA2Rab relative to baseline within 6 months after the first infusion, as well as the overall response rate (CR+PR), complete response rate, partial response rate, and incidence of adverse events related to IM19 CAR-T cell infusion within 28 days after IM19 CAR-T cell infusion.

And evaluate the long-term efficacy, that is, assess the rate of PLA2Rab changes and disappearance relative to baseline, overall response rate (CR+PR), complete response rate, and partial response rate of the subjects after 360 days of cell transfusion. The retention amount and duration of IM19 CAR-T cells in the peripheral blood of subjects.

ELIGIBILITY:
Inclusion Criteria：

* IgA nephropathy

  1. IgA nephropathy diagnosed through renal biopsy
  2. When screening, urine protein should be ≥0.5g/gCr and 20mL/min/1.73m^2≤eGFR<60mL/min/1.73m^2
  3. Age≥18years old
  4. Liver, kidney, heart, lung function, and coagulation function meet the following requirements:

     4.1 ALT and AST ≤ 2.5 × ULN,total bilirubin ≤ 1.5 × ULN (for subjects with Gilbert syndrome, ALT and AST ≤ 5 × ULN, total bilirubin ≤ 3 × ULN); 4.2 Left ventricular ejection fraction ≥ 50%; 4.3 International ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; 4.4 Finger pulse oxygen saturation>92% in non oxygen state;
  5. Women of childbearing age who have a negative blood pregnancy test before the start of the trial and agree to take effective contraceptive measures during the trial period until the last follow-up; Male participants with reproductive partners agree to take effective contraceptive measures during the trial period until the last follow-up;
  6. Doctors evaluate patients with the optimal benefit risk ratio
  7. Those who voluntarily participate in this experiment and sign the informed consent form
* Primary membranous nephropathy:

  1. Diagnosis of primary membranous nephropathy through renal biopsy;
  2. Primary membranous nephropathy at medium or high risk that has not improved after 6 months of treatment with CNI and rituximab:

     2.1. Moderate risk assessment criteria 2.1.1. EGFR is normal, 24-hour urine protein is>4g, and conservative treatment with angiotensin-converting enzyme inhibitors/angiotensin receptor blockers has been continuously used for 6 months or more before screening. The 24-hour urine protein has not decreased by less than 50% 2.1.2. PLA2R antibody<50RU/mL+ 2.1.3. Low molecular weight urinary protein 2.1.4. Selectivity index<0.15 2.1.5. Urinary immunoglobulin UIgG<250mg/day 2.2 High risk assessment criteria 2.2.1. eGFR<60ml/min/1.73m^2 2.2.2. 24-hour urine protein>4g and lasting>6 months 2.2.3. PLA2R antibody>150RU/mL+ 2.2.4. High molecular weight urinary protein 2.2.5. Urine immunoglobulin UigG>250mg/day 2.2.6. Selectivity index>0.20
  3. Age ≥ 18 years old;
  4. Liver, heart, lung function, and coagulation function meet the following requirements:

     4.1. ALT and AST ≤ 2.5 × ULN, total bilirubin ≤ 1.5 × ULN (for) Subjects with Gilbert syndrome, ALT and AST ≤ 5 × ULN, total bilirubin ≤ 3 × ULN); 4.2. Left ventricular ejection fraction ≥ 50%; 4.3. International ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; 4.4. Finger pulse oxygen saturation>92% in non oxygen state
  5. Women of childbearing age who have a negative blood pregnancy test before the start of the trial and agree to take effective contraceptive measures during the trial period until the last follow-up; Male participants with reproductive partners agree to take effective contraceptive measures during the trial period until the last follow-up
  6. Doctors evaluate patients with the optimal benefit risk ratio
  7. Those who voluntarily participate in this experiment and sign the informed consent form

Exclusion Criteria:

* IgA nephropathy:

  1. Kidney diseases other than IgA nephropathy, as well as primary and secondary nephrotic syndrome
  2. After examination by the researchers, it was determined that the subjects had diseases that were not suitable for participation in this study, such as life-threatening conditions (such as catastrophic antiphospholipid syndrome, acute severe renal failure, and acute severe central nervous system disease manifestations)
  3. Serious complications unrelated to IgA nephropathy
  4. Use or increase the dosage of corticosteroids, immunosuppressants, biologics (including but not limited to CD20 monoclonal antibodies, taceptil, etc.), anticoagulants (warfarin), and n-3 fatty acids (fish oil) for the drug treatment of IgA nephropathy within 3 months
  5. Uncontrollable hypertension or hyperglycemia
  6. Perform palatal tonsillectomy within 6 months
  7. Study subjects with a history of alcohol or drug abuse within the past 24 weeks
  8. Have undergone major surgery (including joint surgery) within 24 weeks prior to screening, or plan to undergo surgery within 24 weeks after enrollment in the study
  9. Used other cell therapies
  10. Have participated in or participated in other clinical trials within the past 3 months
  11. Within 3 years or planning to undergo a kidney transplan
  12. Active hepatitis B or hepatitis C virus, defined as: subjects with positive hepatitis B B virus surface antigen (HBsAg) and/or hepatitis B B core antibody (HBcAb, Hepatitis B core antibody) and HBV DNA titer in peripheral blood higher than the lower limit of detection; Individuals with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA (HCV RNA); Syphilis infected individuals
  13. Active EB virus and cytomegalovirus, defined as: subjects with positive or negative IgM antibodies in EB virus serum but EBV-DNA higher than normal values; Subjects with IgM antibody positive or IgM antibody negative but CMV-DNA higher than normal in the serum of cytomegalovirus (CMV)
  14. Serious history of cardiovascular and cerebrovascular diseases, including but not limited to:

      14.1. Serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, third degree atrioventricular block, etc; 14.2. At rest, QT interval prolongation (QTc>450 milliseconds in males or>470 milliseconds in females); 14.3. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months prior to the first administration; 14.4. There is heart failure with NYHA functional class ≥ II in the United States;
  15. History of symptomatic deep vein thrombosis or pulmonary embolism within the past 6 months prior to the start of screening;
  16. History of malignant tumors other than non melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) (unless in a disease-free state for at least 3 years)
  17. Infections (fungal, bacterial, viral, or other) that require intravenous injection of antibiotics for control or are uncontrollable, such as simple urinary tract infections and bacterial pharyngitis, may be included if the researcher evaluates that they can be controlled through treatment
  18. The researchers believe that it does not meet the criteria for joining this clinical trial
  19. During pregnancy or lactation, it may be due to pregnancy or the male and female not agreeing to undergo contraception under the guidance of the researcher during the study period.
* Primary membranous nephropathy:

  1. Secondary membranous nephropathy;
  2. Urinary protein decreased by more than 50% within the first 6 months of screening;
  3. After examination by the researchers, it was determined that the subjects had diseases that were not suitable for participation in this study, such as life-threatening conditions (such as catastrophic antiphospholipid syndrome, acute severe renal failure, and acute severe central nervous system disease manifestations);
  4. Serious complications unrelated to primary membranous nephropathy;
  5. Uncontrollable hypertension or hyperglycemia;
  6. The study subjects have a history of alcohol or drug abuse within the past 24 weeks;
  7. Have undergone major surgery (including joint surgery) within 24 weeks prior to screening, or plan to undergo surgery within 24 weeks after enrollment in the study;
  8. Have used other cell therapies;
  9. Have participated in or taken part in other clinical trials within the past 3 months;
  10. Within 3 years or planning to undergo kidney transplantation;
  11. Active hepatitis B or hepatitis C virus, defined as: subjects with positive hepatitis B B virus surface antigen (HBsAg) and/or hepatitis B B core antibody (HBcAb, Hepatitis B core antibody) and HBV DNA titer in peripheral blood higher than the lower limit of detection; Individuals with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA (HCV RNA); Syphilis infected individuals;
  12. Active EB virus and cytomegalovirus, defined as: subjects with positive or negative IgM antibodies in EB virus serum but EBV-DNA higher than normal values; Subjects with IgM antibody positive or IgM antibody negative but CMV-DNA higher than normal in the serum of cytomegalovirus (CMV);
  13. History of serious cardiovascular and cerebrovascular diseases, including but not limited to: severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, third degree atrioventricular block, etc; At rest, QT interval prolongation (QTc>450 milliseconds in males or>470 milliseconds in females); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months prior to the first administration; There is heart failure with NYHA functional class ≥ II in the United States;
  14. History of symptomatic deep vein thrombosis or pulmonary embolism within the past 6 months prior to the start of screening;
  15. History of malignant tumors other than non melanoma skin cancer or carcinoma in situ (such as cervix, bladder, breast) (unless in a disease-free state for at least 3 years);
  16. Infections (fungal, bacterial, viral, or other) that require intravenous injection of antibiotics for control or are uncontrollable, such as simple urinary tract infections and bacterial pharyngitis, may be included if the researcher evaluates that they can be controlled through treatment;
  17. The researcher believes that it does not meet the criteria for joining this clinical trial;
  18. During pregnancy or lactation, it may be due to pregnancy or the male and female not agreeing to undergo contraception under the guidance of the researcher during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-13 (Estimated); Primary Completion 2025-08-04 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
IgA nephropathy-Main safety endpoint（Adverse event incidence rate） | IM19 CAR-T cell reinfusion within 28 days
  The incidence of adverse events related to IM19 CAR-T cell reinfusion within 28 days after IM19 CAR-T cell reinfusion, as well as clinically significant laboratory test results.
IgA primary efficacy endpoint（Urinary protein ratio） | 6 months after the first administration
  Changes in urinary protein levels (1 day, 14 days, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months after initial administration) relative to baseline values and the rate of reaching the threshold
PMN primary safety endpoint（Adverse event incidence rate） | IM19 CAR-T cell reinfusion within 28 days
  The incidence of adverse events related to IM19 CAR-T cell reinfusion within 28 days after IM19 CAR-T cell reinfusion, as well as clinically significant laboratory test results.
PMN primary efficacy endpoint（Relief rate） | 6 months after the first administration
  Evaluate the overall response rate (CR+PR), complete response rate, and partial response rate of the subjects 6 months after the first infusion.
  Complete remission criteria: Urinary protein ≤ 0.3g and serum albumin>3.5g/dl. Partial relief criteria: Urinary protein reduction>50% compared to baseline and final 0.3g<urinary protein ≤ 3.5g.

SECONDARY OUTCOMES:
IgA secondary endpoint（EGFR ratio） | 360 days after IM19 CAR-T cell reinfusion
  The ratio of eGFR levels reaching the threshold after IM19CAR-T cell reinfusion
IgA secondary endpoint（Urinary protein ratio） | 360 days after IM19 CAR-T cell reinfusion
  The ratio of urinary protein levels reaching the threshold after IM19CAR-T cell reinfusion
PMN secondary endpoint（Relief rate） | 360 days after IM19 CAR-T cell reinfusion
  Evaluate the rate of relative baseline changes and disappearance of PLA2Rab, overall response rate (CR+PR), complete response rate, and partial response rate in subjects after 360 days of cell transfusion

CONTACTS AND LOCATIONS:
Overall Officials: xiangmei Chen, doctorate, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No